CLINICAL TRIAL: NCT05683665
Title: DaTSCAN Brain Scintigraphy and Psychotropic Treatments: Influence on Radiotracer Binding
Acronym: DAPSYFIX
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2022PI098
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: scintigraphy DaTSCAN — DaTSCAN™ (123I-ioflupnae) tomoscintigraphy assesses the density of dopamine transporters (DATs) on the pre-synaptic membrane of dopaminergic neurons

SUMMARY:
DaTSCAN™ (123I-ioflupnae) tomoscintigraphy assesses the density of dopamine transporters (DATs) on the presynaptic membrane of dopaminergic neurons. This examination is used in clinical routine in patients presenting a parkinsonian syndrome in search of a pre-synaptic dopaminergic denervation pointing to a neurodegenerative origin of this syndrome To date, there is little literature data evaluating the influence of psychotropic treatments frequently used in clinical routine on DaTSCAN™ CT images. Some studies have shown that SSRI (selective serotonin reuptake inhibitor) and SNRI (serotonin and norepinephrine reuptake inhibitor) antidepressants can significantly alter striatal ioflupane uptake ratios (10-20%) with no obvious influence on the visual interpretation of the examination .

The objective of this study was to evaluate the influence of the most commonly used psychotropic therapies, sometimes in combination, on DaTSCAN™ CT images with a large population of patients included in clinical routine.

DETAILED DESCRIPTION:
DaTSCAN™ (123I-ioflupnae) tomoscintigraphy assesses the density of dopamine transporters (DATs) on the presynaptic membrane of dopaminergic neurons. This examination is used in clinical routine in patients presenting a parkinsonian syndrome in search of a pre-synaptic dopaminergic denervation pointing to a neurodegenerative origin of this syndrome Some drugs, and in particular psychotropic treatments, have an ability to bind to dopamine transporters or to mobilize endogenous dopamine and may thus interfere with ioflupane binding. Visual interpretation of the DaTSCAN™ scan as well as semi-quantitative analysis (radiotracer binding ratios) takes into account striatal binding activity and also activity in the rest of the brain parenchyma (background) . Therefore, drugs that interfere with striatal or extra-striatal binding of ioflupane may have an impact on the examination result.

To date, there is little literature data evaluating the influence of psychotropic treatments frequently used in clinical routine on DaTSCAN™ CT images. Some studies have shown that SSRI (selective serotonin reuptake inhibitor) and SNRI (serotonin and norepinephrine reuptake inhibitor) antidepressants can significantly alter striatal ioflupane uptake ratios (10-20%) with no obvious influence on the visual interpretation of the examination . Antipsychotic and antiparkinsonian drugs appear to have no effect on ioflupane uptake and should not be discontinued before the examination is performed. Finally, lithium treatment could significantly reduce ioflupane binding.

The majority of studies analyzing the effects of medication on ioflupane binding have been conducted in small numbers or assess the potential impact of therapy on a theoretical basis.

The objective of this study was to evaluate the influence of the most commonly used psychotropic therapies, sometimes in combination, on DaTSCAN™ CT images with a large population of patients included in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson syndroma
* Patients with Datscan in Nancy hospital bewteen septemnre 2019 and december 2022

Exclusion Criteria:

* Patient with a known allergy to any of the components of DaTSCAN™.
* Patient deprived of liberty by a judicial or administrative decision

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients routinely referred for SPECT examination assessing the pre-synaptic dopaminergic pathway
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The influence of psychotropic treatments on radiotracer uptake during DaTSCAN™ tomoscintigraphies. | 1 year
  Binding ratios (specific binding ratio) stratum/occipital cortex, caudate nucleus/occipital cortex, putamen/occipital cortex on the left and right and total number of strokes recorded as a function of the presence or absence of psychotropic treatment at the time of examination

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France